CLINICAL TRIAL: NCT02836223
Title: Evaluation of the Addition of an Interdental Cleaning Device to Manual Brushing on Gingival Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Water Pik, Inc. (Industry)
Collaborators: All Sum Research Center Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16WFVSMTB2016
Record Dates: First submitted 2016-07-14; First posted 2016-07-18 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-07

CONDITIONS: Gingivitis
MeSH Terms: conditions — Gingivitis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Interdental device (Experimental): Water Flosser
  Interventions: Device: Interdental cleaning device; Device: Manual Tooth brush
- Toothbrush (Other): Control
  Interventions: Device: Manual Tooth brush

INTERVENTIONS:
Device: Interdental cleaning device — Water Flosser
  Arms: Interdental device
Device: Manual Tooth brush — Control

SUMMARY:
This study evaluates the addition of an interdental cleaning device paired with a manual toothbrush compared to using a manual toothbrush only. Plaque removal, reduction of gingival bleeding and reduction of gingival inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Between 25 and 70 years of age
* Able to provide written informed consent prior to participation
* Agree to not participate in any other oral/dental products clinical study for the study duration
* Good general health and be a non-smoker
* A minimum of 50% bleeding on probing sites
* A minimum pre-brushing plaque score of 0.6
* A minimum of 1.75 gingivitis score Have no probing depths greater than 5 mm
* A minimum of 20 teeth (not including 3rd molars)
* No partial dentures, orthodontic brackets, wires or other appliances
* Agree to refrain from the use of any non-study dental device or oral care product for the study duration
* Agree to return for the scheduled visits and follow study procedures
* Agree to delay dental prophylaxis until study completion
* Have a minimum pre-brushing plaque score of 0.6
* Have a minimum of 1.75 gingivitis score

Exclusion Criteria:

* Probing depth greater than 5 mm
* Systemic disease (ex. Diabetes, autoimmune disease)
* Advanced periodontitis
* Taking medication that can influence gingival health such as seizure meds, calcium channel blockers, Cyclosporine, anticoagulants
* Orthodontic appliances or removable partial dentures
* Pregnant at time of study
* Use of antibiotics within 6 months of study

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2016-07; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Reduction of gingival bleeding | 4 weeks

SECONDARY OUTCOMES:
Reduction of gingival inflammation | 4 weeks
Reduction in dental plaque | 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- All Sum Research Center Ltd., Mississauga, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No